CLINICAL TRIAL: NCT01925716
Title: A Randomized Double Blind Controlled Crossover Trial to Assess the Effects of Dietary Oils on Fasting Lipoprotein Lipids
Brief Title: Effects of The Effects of Dietary Oils on Fasting Lipoprotein Lipids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ACH Food Companies, Inc. (Industry)
Collaborators: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: PRV-1303
Record Dates: First submitted 2013-08-14; First posted 2013-08-20 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Hypercholesterolemia
Keywords: cholesterol,LDL; vegetable oils; heart diseases
MeSH Terms: conditions — Hypercholesterolemia; Heart Diseases | interventions — Corn Oil; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corn oil/olive oil (Experimental): Corn oil 56 g per day for 21 days followed by olive oil 56 g for 21 days
  Interventions: Other: Corn oil; Other: Olive oil
- Olive Oil/Corn Oil (Experimental): olive oil, 56g per day for 21 days followed by corn oil, 56 g for 21 days
  Interventions: Other: Corn oil; Other: Olive oil

INTERVENTIONS:
Other: Corn oil — corn oil 56 g/day for 21 days
Other: Olive oil — olive oil 56 g /day for 21 days

SUMMARY:
The objectives of this clinical trial are to assess the effects of dietary oils on blood lipids and other aspects of the fasting lipoprotein profile in healthy men and women with elevated cholesterol

ELIGIBILITY:
Inclusion Criteria:

* Fasting LDL-C level equal to or greater than 130 mg/dL and less than 200 mg/dL at visit 1
* Fasting triglycerides less than or equal to 350 mg/dL at visit 1

Exclusion Criteria:

* Has coronary heart disease or coronary heart disease risk risk equivalent, such as diabetes, atherosclerosis, etc
* Taking lipid medications intended to alter the lipids profile, including but not limited to statins, bile acid sequestrants, etc.
* Uncontrolled hypertension (systolic greater than or equal to 160 mm Hg or diastolic greater than or equal to 100 mm Hg)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Low Density Lipoprotein cholesterol | Time Frame: baseline (average days -7 and 0) and the end of each treatment period [Treatment 1 averages of days 19 and 21and Treatment II (average of days 19 and 21)]: patients are followed for an average of 11 weeks

SECONDARY OUTCOMES:
total cholesterol | baseline (average of days -7 and 0) and the end of each treatment period [Treatment I average of days 19 and 21) and treatment II (average of days 19 and 21)]: patients are followed for an average of 11 weeks

OTHER OUTCOMES:
High density lipoprotein cholesterol | baseline (average of days -7 and 0) and the end of each treatment period [Treatment I average of days 19 and 21) and treatment II (average of days 19 and 21)]: patients are followed for an average of 11 weeks
Non-HDL-Cholesterol | baseline (average of days -7 and 0) and the end of each treatment period [Treatment I average of days 19 and 21) and Treatment II (average of days 19 and 21)]: patients are followed for an average of 11 weeks
Triglycerides | baseline (average of days -7 and 0) and the end of each treatment period [Treatment I average of days 19 and 21) and Treatment II (average of days 19 and 21)]: patients are followed for an average of 11 weeks
Total cholesterol/HDL-C ratio | baseline (average of days -7 and 0) and the end of each treatment period [Treatment I average of days 19 and 21) and Treatment II (average of days 19 and 21)]: patients are followed for an average of 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Maki, PhD, Study Director — Biofortis Clinical Research, Inc.

REFERENCES:
- [Derived] Maki KC, Lawless AL, Kelley KM, Kaden VN, Geiger CJ, Dicklin MR. Corn oil improves the plasma lipoprotein lipid profile compared with extra-virgin olive oil consumption in men and women with elevated cholesterol: results from a randomized controlled feeding trial. J Clin Lipidol. 2015 Jan-Feb;9(1):49-57. doi: 10.1016/j.jacl.2014.10.006. Epub 2014 Oct 23. PMID 25670360